CLINICAL TRIAL: NCT05045326
Title: Effectiveness of a Smoking Cessation Intervention in a Mental Health Day Hospital
Acronym: ESCIM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HCB/2019/0580
Record Dates: First submitted 2021-07-29; First posted 2021-09-16 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Tobacco Use Disorder; Smoking Cessation; Mental Disorder
Keywords: Motivational Interviewing; Group Counseling
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Intervention Group (Experimental): Participants in the intervention group will receive an intensive motivational intervention with individual and group treatment for smoking cessation. The treatment, provided by trained professionals, will include psychological, psycho-educational support and pharmacological treatment advice.
  Interventions: Behavioral: Smoking cessation program
- Placebo Comparator: Brief Counselling (Placebo Comparator): Participants in the placebo group will receive a brief intervention for smoking cessation.
  Interventions: Behavioral: Placebo Comparator: Brief Counselling

INTERVENTIONS:
Behavioral: Smoking cessation program — Participants will receive intensive treatment for smoking cessation during day hospital admission.
  The intervention is carried out individually and in an open-ended group. The treatment, provided by trained and multidisciplinary professionals (nursing, psychiatry, psychologist, occupational therapist, social work), includes psychological, psycho-educational support, and pharmacological treatment advice.
  The group intervention takes place once a week and is divided into six structured sessions that are repeated. Sessions include nicotine addiction and withdrawal, health consequences, benefits of quitting, motivation for change, triggers, coping responses, social support, decision making, pharmacological treatment advice and healthy lifestyle habits.
  Arms: Experimental: Intervention Group
Behavioral: Placebo Comparator: Brief Counselling — Participants will receive brief counseling on smoking cessation during their hospital stay. This brief intervention is based on motivational techniques to increase motivation to reduce tobacco use or to initiate treatment.
  Arms: Placebo Comparator: Brief Counselling

SUMMARY:
Background: Nicotine contained in tobacco is highly addictive and tobacco use is a major risk factor for cardiovascular and respiratory diseases. Every year, more than 8 million people die from tobacco use.

Smoking-related mortality is significantly higher in people with serious mental illness. Is estimated that half of all deaths among individuals with mental illnesses are attributable to tobacco use. People with serious mental illness have greater daily tobacco consumption, nicotine dependence, and smoking relapse. While significant progress has been made in reducing tobacco use within the general population, rates of tobacco use remain high among individuals with mental illness. Smoking cessation often requires numerous attempts by these people. Thus, smokers with mental health illnesses may find it more difficult to quit, although highly motivated to quit.

Smoking cessation during hospitalization (total or partial) is cost-effective, as it reduces hospital readmissions, and mortality, and improves smokers' quality of life. Available quitting aids are both safe and effective in supporting cessation in tobacco users with mental illness and stopping smoking is associated with an improvement in mental health.

The investigators aimed to evaluate the feasibility and efficacy of adding an intensive smoking intervention to the usual treatment for patients with psychiatric disorders attending a day hospital of a tertiary hospital.

DETAILED DESCRIPTION:
The investigators will perform a quasi-experimental, longitudinal, and prospective study in the mental health day hospital of the Hospital Clinic of Barcelona.

Adults attending the day hospital and willing to participate, under informed consent, will be invited to participate. Consecutive eligible individuals will be recruited and will be assigned to two groups, the control group, and the experimental group. Initially, patients will be recruited for the control group, once the control group is completed the experimental group will begin.

An assessment will be conducted at baseline (admission) and in the discharge. Sociodemographic and clinical data will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Mental health day hospital inpatient.
* Smoker of at least 1 cigarette per day, electronic cigarette, or heated tobacco product daily for at least 1 month.
* Individuals who accept to participate in the study and give informed consent.

Exclusion Criteria:

* Cognitive impairment, dementia, or brain damage.
* Medically unstable.
* Explicitly demanding tobacco treatment.
* Trying to quit smoking using another intervention.
* Insufficient comprehension skills in Spanish or Catalan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-05-30 (Actual); Primary Completion 2023-07-27 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Tobacco use changes from baseline to post-intervention | An average of 2 months
  Number of cigarettes smoked in past 24 hours.
Motivation to quit smoking changes from baseline to post-intervention | An average of 2 months
  Individuals will be assessed with the Richmond test.
Cotinine levels in urine changes from baseline to post-intervention | An average of 2 months
  Urine cotinine levels

SECONDARY OUTCOMES:
Nicotine dependence changes from baseline to post-intervention | An average of 2 months
  Change of self reported tobacco dependence using Fagerström Test for Nicotine Dependence.
Self-efficacy to quit smoking changes from baseline to post-intervention | An average of 2 months
  Change of self reported self-efficacy (using a Likert scale from 0 to 10). Minimum value: 0. Maximum value: 10. Higher scores indicate more self-efficacy to quit smoking.
Smoking knowledge changes from baseline to post-intervention | An average of 2 months
  Changes in smoking knowledge obtained through a knowledge questionnaire developed by the researchers.
Trait and state anxiety changes from baseline to post-intervention | An average of 2 months
  Changes in anxiety obtained through the State-Trait Anxiety Inventory. Minimum value: 20. Maximum value: 80. Higher scores indicate greater anxiety.
Depressive symptoms changes from baseline to post-intervention | An average of 2 months
  Changes in depressive symptoms obtained through the Montgomery and Asberg Depression. Minimum value: 0 Maximum value: 60. A score of less than 10 points indicate the absence of depressive disorder.
Self-reported clinically relevant psychological symptoms changes from baseline to post-intervention | An average of 2 months
  Changes in self-reported clinically relevant psychological symptoms through the Brief Symptom Inventory. Minimum value: 0. Maximum value: 72. Higher scores indicate higher levels of psychological distress.

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Gual, PhD, MD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rogers ES, Gillespie C, Smelson D, Sherman SE. A Qualitative Evaluation of Mental Health Clinic Staff Perceptions of Barriers and Facilitators to Treating Tobacco Use. Nicotine Tob Res. 2018 Sep 4;20(10):1223-1230. doi: 10.1093/ntr/ntx204. PMID 29059344
- [Background] Japuntich SJ, Hammett PJ, Rogers ES, Fu S, Burgess DJ, El Shahawy O, Melzer AC, Noorbaloochi S, Krebs P, Sherman SE. Effectiveness of Proactive Tobacco Cessation Treatment Outreach Among Smokers With Serious Mental Illness. Nicotine Tob Res. 2020 Aug 24;22(9):1433-1438. doi: 10.1093/ntr/ntaa013. PMID 31957794
- [Background] Martin-Cantera C, Sanmartin JMI, Martinez AF, Lorenzo CM, Cohen VB, Jimenez MLC, Perez-Teijon SC, Osca JARI, Garcia RC, Fernandez JL, Domenech MAG, Navascues MAM, Chaves ES, Ibanez MLR, Rubio VG, Rayo SM, Otero BM, Lopez LG, Guillem FC, Fuente FM, Ruiz DB, Rodriguez AIH, Caballero JDG, Moreno CB, Pubil MP, Grau ML. Good practice regarding smoking cessation management in Spain: Challenges and opportunities for primary care physicians and nurses. Tob Prev Cessat. 2020 Sep 21;6:55. doi: 10.18332/tpc/126630. eCollection 2020. PMID 33083683
- [Background] Godoy R, Callejas FJ, Cruz J, Tornero AI, Tarraga PJ, Rodriguez-Montes JA. [Comparative analysis: Effectiveness of nicotine addiction treatment in people with psychiatric comorbidity]. Semergen. 2018 May-Jun;44(4):249-256. doi: 10.1016/j.semerg.2017.03.008. Epub 2017 Jun 20. Spanish. PMID 28645694
- [Background] Rice VH, Heath L, Livingstone-Banks J, Hartmann-Boyce J. Nursing interventions for smoking cessation. Cochrane Database Syst Rev. 2017 Dec 15;12(12):CD001188. doi: 10.1002/14651858.CD001188.pub5. PMID 29243221
- [Background] Lindson N, Thompson TP, Ferrey A, Lambert JD, Aveyard P. Motivational interviewing for smoking cessation. Cochrane Database Syst Rev. 2019 Jul 31;7(7):CD006936. doi: 10.1002/14651858.CD006936.pub4. PMID 31425622
- [Background] Jaen-Moreno MJ, Feu N, Redondo-Ecija J, Montiel FJ, Gomez C, Del Pozo GI, Alcala JA, Gutierrez-Rojas L, Balanza-Martinez V, Chauca GM, Carrion L, Osuna MI, Sanchez MD, Caro I, Ayora M, Valdivia F, Lopez MS, Poyato JM, Sarramea F. Smoking cessation opportunities in severe mental illness (tobacco intensive motivational and estimate risk - TIMER-): study protocol for a randomized controlled trial. Trials. 2019 Jan 14;20(1):47. doi: 10.1186/s13063-018-3139-9. PMID 30642365
- [Background] Jordan K. A Provider - Patient Relationship: The Critical First Step of Smoking Cessation. J Gen Intern Med. 2020 Jan;35(1):10-11. doi: 10.1007/s11606-019-05276-0. No abstract available. PMID 31720963
- [Background] Guydish J, Wahleithner J, Williams D, Yip D. Tobacco-free grounds implementation in California residential substance use disorder (SUD) treatment programs. J Addict Dis. 2020 Jan-Mar;38(1):55-63. doi: 10.1080/10550887.2020.1713687. Epub 2020 Jan 25. PMID 32186480
- [Background] Knudsen HK. Implementation of smoking cessation treatment in substance use disorder treatment settings: a review. Am J Drug Alcohol Abuse. 2017 Mar;43(2):215-225. doi: 10.1080/00952990.2016.1183019. Epub 2016 Jun 17. PMID 27314884
- [Background] Malone V, Harrison R, Daker-White G. Mental health service user and staff perspectives on tobacco addiction and smoking cessation: A meta-synthesis of published qualitative studies. J Psychiatr Ment Health Nurs. 2018 May;25(4):270-282. doi: 10.1111/jpm.12458. Epub 2018 Apr 14. PMID 29498459
- [Background] Martinez C, Castellano Y, Andres A, Fu M, Feliu A, Anton L, Ballbe M, Fernandez P, Cabrera S, Riccobene A, Gavilan E, Baena A, Margalef M, Tigova O, Quiros N, Guillen O, Company A, Fernandez E. Impact of an Online Training Program in Smoking Cessation Interventions in Hospitals. J Nurs Scholarsh. 2019 Jul;51(4):449-458. doi: 10.1111/jnu.12469. Epub 2019 Mar 15. PMID 30874373
- [Background] Martinez C, Feliu A, Castellano Y, Fu M, Fernandez P, Cabrera-Jaime S, Puig-Llobet M, Galimany J, Guydish J, Fernandez E; ETHIF Research Group. Factors associated with receipt of the 5As model of brief intervention for smoking cessation among hospitalized patients. Addiction. 2020 Nov;115(11):2098-2112. doi: 10.1111/add.15076. Epub 2020 Apr 28. PMID 32297373
- [Background] Andres A, Castellano Y, Fu M, Feliu A, Ballbe M, Anton L, Baena A, Fernandez E, Martinez C. Exploring individual and contextual factors contributing to tobacco cessation intervention implementation. Addict Behav. 2019 Jan;88:163-168. doi: 10.1016/j.addbeh.2018.08.003. Epub 2018 Aug 6. PMID 30205255
- [Background] Peckham E, Brabyn S, Cook L, Tew G, Gilbody S. Smoking cessation in severe mental ill health: what works? an updated systematic review and meta-analysis. BMC Psychiatry. 2017 Jul 14;17(1):252. doi: 10.1186/s12888-017-1419-7. PMID 28705244
- [Background] Muller DP, de Haan L. [Smoking cessation and schizophrenia]. Tijdschr Psychiatr. 2017;59(5):297-301. Dutch. PMID 28593623
- [Background] Zvolensky MJ, Rosenfield D, Garey L, Kauffman BY, Langdon KJ, Powers MB, Otto MW, Davis ML, Marcus BH, Church TS, Frierson GM, Hopkins LB, Paulus DJ, Baird SO, Smits JAJ. Does exercise aid smoking cessation through reductions in anxiety sensitivity and dysphoria? Health Psychol. 2018 Jul;37(7):647-657. doi: 10.1037/hea0000588. Epub 2018 Apr 30. PMID 29708388
- [Background] Nieva G, Ballbe M, Cano M, Carcole B, Fernandez T, Martinez A, Mondon S, Raich A, Roig P, Serra I, Serrano J, Pinet C. Smoking cessation interventions in substance use disorders treatment centers of Catalonia: The abandoned addiction. Adicciones. 2022 Jul 1;34(3):227-234. doi: 10.20882/adicciones.1492. English, Spanish. PMID 33768256
- [Background] Healey A, Roberts S, Sevdalis N, Goulding L, Wilson S, Shaw K, Jolley C, Robson D. A Cost-Effectiveness Analysis of Stop Smoking Interventions in Substance-Use Disorder Populations. Nicotine Tob Res. 2019 Apr 17;21(5):623-630. doi: 10.1093/ntr/nty087. PMID 29733376
- [Background] Ballbe M, Gual A, Nieva G, Salto E, Fernandez E; Tobacco and Mental Health Working Group. Deconstructing myths, building alliances: a networking model to enhance tobacco control in hospital mental health settings. Gac Sanit. 2016 Sep-Oct;30(5):389-92. doi: 10.1016/j.gaceta.2016.04.017. Epub 2016 Jun 17. PMID 27325123
- See also: The World Health Organization report on the global tobacco epidemic 2019: offer help to quit tobacco use" tracks the status of the tobacco epidemic and interventions to combat it. — https://www.who.int/teams/health-promotion/tobacco-control/who-report-on-the-global-tobacco-epidemic-2019
- See also: Clinical Intervention guide on tobacco use in patients with mental disorders. Government of Catalonia. 2012. — https://www.xchsf.cat/docs/460-Guia%20Tabac%20int%20cast.pdf